CLINICAL TRIAL: NCT01122641
Title: Does Modulating the Gut Hormones, Incretins, Modify Vascular Function, Thereby Reducing the Risk of Vascular Complications in Insulin Resistant Individuals?
Brief Title: The Vascular Effects of Vildagliptin in Insulin Resistant Individuals
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, David Strain, PI, Royal Devon and Exeter NHS Foundation Trust
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 2009-013100-32; 09/H0206/33 (Other: REC study number)
Record Dates: First submitted 2010-05-12; First posted 2010-05-13 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Insulin Resistance; Microvascular Disease
Keywords: Insulin resistance; incretins; DPP4 inhibitors; vildagliptin; microcirculation
MeSH Terms: conditions — Insulin Resistance | interventions — Vildagliptin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Vildagliptin (Experimental): Vildagliptin 50mg bid
  Interventions: Drug: Vildagliptin

INTERVENTIONS:
Drug: Vildagliptin — Vildagliptin 50mg bid
  Other Names: Galvus
  Arms: Vildagliptin
Drug: Placebo — Matched tablets
  Arms: Placebo

SUMMARY:
Animal models have demonstrated that incretins have a glucose-independent effect on vascular perfusion, and there is limited evidence that incretins may enhance endothelial function in healthy subjects. Currently DPP-4 inhibition increases levels of the endogenous incretin Glucagon-like Peptide 1 (GLP-1) and is licensed for the treatment of hyperglycaemia in type 2 diabetes. They are positioned as third or even fourth line therapy after metformin, sulphonylureas ± glitazones, however recent analyses of cardiovascular outcomes in glitazones and sulphonylureas suggest at best they do not reduce cardiovascular endpoints, and may increase some outcomes. If the vascular benefits suggested in animal models are realised in humans this should see the DPP-4 inhibitors moved to second line and possibly 1st line.

In order to realise the potential the investigators would like initially to demonstrate increases in vascular perfusion and function in a placebo controlled trial using accurate surrogates for vascular function in patients with insulin resistance and obesity.

The investigators hypothesis is that by increasing incretin activity in insulin resistant states the investigators will lower capillary pressure and improve microvascular function, which will be accompanied by a reduction in macular thickness (by reducing macular oedema) and microalbuminuria, recognised surrogates for early diabetic retinopathy and renal failure respectively.

DETAILED DESCRIPTION:
After food intake, insulin secretion depends not only on the degree of glycemia, but also on the secretion and insulinotropic effect of the gut hormones, gastric inhibitory polypeptide (or glucose-dependent insulinotropic polypeptide; GIP) and glucagon-like polypeptide 1 (GLP-1), known as incretins. Normally, the incretins GLP-1 and GIP are responsible for as much as half of the glucose-dependent insulin release after food ingestion. In obesity and patients with insulin resistance the GIP and GLP-1 responses to a mixed meal are impaired and in the latter case are related to the degree of insulin resistance[1, 2]. In subjects with type 2 diabetes, the insulin releasing action of GIP is reduced, however GLP-1 responsiveness is normal [3]. This has resulted in the successful use of therapies either increasing endogenous GLP-1 (by inhibiting its breakdown by dipeptidyl-peptidase IV; DPP-IV) or administering synthetic GLP-1 in order to treat the hyperglycaemia of type 2 diabetes. It is widely recognised, however, that diabetes and insulin resistance adversely impacts vascular function, independently of hyperglycaemia, resulting in premature ischaemic heart disease, stroke, retinopathy leading to blindness, renal failure and peripheral vascular disease.

Dysfunction of the vasculature, both in macro- and microcirculation, is well described in people with diabetes. Further, altered vascular function has been demonstrated in individuals predisposed to diabetes, for example in subjects with fasting hyperglycaemia [4], impaired glucose tolerance [5], in women with previous gestational diabetes [6], in obese individuals [7, 8] and in 3 month old infants of low birth weight [9]. Unpublished data from our own laboratory demonstrates capillary pressure is positively associated with fovea (macular) thickness, the thickening of which is an early pre-clinical sign of macular oedema, in healthy subjects with a wide range of body mass index (BMI) that varies from the lean to the morbidly obese (20.0 - 46.6 m2/kg). In patients with established retinopathy treatments that reduce fovea thickness are associated with improvements of visual acuity, whereas increasing fovea thickness was associated with a trend towards poorer eyesight [10].

Microangiopathy appears to precede the development of cardiovascular events in those with diabetes [11], and changes in microvascular function appear to precede this microangiopathy [12, 13]. Therapies that improve clinically detectable evidence of microangiopathy, such as microalbuminuria, have demonstrated improvements in cardiovascular outcomes independent of their antihypertensive effect [14-16]. In the latter of these studies there was a linear relationship between reduction in albumin excretion rate and cardiovascular outcome that was independent of the intervention suggesting that microangiopathy is integral to the aetiopathogenesis of cardiovascular disease. Thus it may be possible that by improving vascular function, for example lowering capillary pressure, we may be able to prevent or delay the progression of clinical vascular complications (eg macular oedema and increased risk of cardiovascular disease) in individuals with or at risk of diabetes. In these cases the administration of therapy that improves both glycaemic control and vascular function will be of enormous health benefit.

There is growing evidence that GLP-1 may have such favourable effects on vascular function, independent of its glucose lowering effects. GLP-1 administration in animal models has been shown to mediate endothelial dependent relaxation in the rat pulmonary artery [17, 18], which was attenuated in the presence of a nitric oxide synthase blocker suggesting the involvement of nitric oxide (NO) in mediating its vascular effects. This is supported by observations that GLP-1 promotes NO-dependent relaxation of mouse mesenteric arteries [19]. This does vary by vascular bed, causing endothelial independent relaxation, via the GLP-1 receptor, in femoral arteries [20] but has no impact on rat aorta isolates [17]. GLP-1 is also protective against ischaemia-reperfusion injury in isolated rat hearts [19, 21-24] and has renoprotective (reducing proteinuria and microalbuminuria) effects, in addition, to the cardio protective effects in Dahl salt sensitive hypertensive rats [25]. Whether these effects are mediated directly via the GLP-1 receptor is unclear, as the vasodilatory effects have been observed to be both dependent[20] and independent [19] of the GLP-1 receptor. In the latter of these studies GLP-1(9-36), which is the product from the degradation of GLP-1 by dipeptidyl peptidase-IV (DPP-IV), mediated relaxation of mouse mesenteric arteries [19]. Thus it is clearly evident that GLP-1 acts as a vasodilator and has cardio protective properties.

Work in humans is still at a more embryonic stage, although the literature looks similarly promising. Acute administration of GLP-1 increases flow mediated dilatation (endothelial dependent) in type 2 diabetic male subjects with coronary artery disease but had no significant effect on young healthy, lean male subjects[26]. In a broader general population sample aged 18-50, GLP-1 does improve forearm blood flow (approx 30% increase) and augments endothelial dependent forearm blood flow response to acetylcholine (approx 40% increase) [27]. Conversely, endothelial independent function is not influenced by the acute administration of GLP-1 in either diabetic or healthy individuals [26, 27]. GLP-1 infusions have also been shown to improve regional and global left ventricular function when administered within 6 hours of an acute myocardial infarction and improve systolic function after successful primary angioplasty in those with severe left ventricular dysfunction [28].

Much work has been completed using direct administration of a GLP-1 mimetic, however, in clinical practice, patient tolerability of repeated subcutaneous injections limits utilisation in the early stages of diabetes. There is little work to date exploring the role of DPP-IV inhibition on vascular function. It is reasonable to assume that the effects of DPP-IV inhibitors (the "gliptins") will not be as impressive as direct GLP-1 administration, as lower levels of GLP-1 are achieved, however longer term therapy is more tolerable and acceptable, due to their simple oral administration and good side-effect profile. It is crucial, therefore, to determine whether these agents prompt clinically relevant improvements in vascular function and thereby attenuate the inevitable cardiovascular decline observed in insulin resistance, and this would necessarily alter current prescribing pathways and guidelines.

Study Question

This study aims to explore the effects of the DPP-IV inhibitor, vildagliptin, on a range of macro- and microvascular parameters. Specific hypotheses to be tested include:

1. increased incretin activity by administration of the DPP-IV inhibitor vildagliptin will lower capillary pressure and improve microvascular function (skin maximum microvascular blood flow, endothelial dependent and independent function) in insulin resistant individuals.
2. improved microvascular function will which will be accompanied by a reduction in macular thickness (by reducing macular oedema) and microalbuminuria, recognised surrogates for early diabetic retinopathy and renal failure respectively.
3. administration of vildagliptin will improve macrovascular function (flow mediated dilatation and arterial stiffness) in insulin resistant individuals.

ELIGIBILITY:
Inclusion Criteria:

* Obese (BMI >30)
* High FinRisk score

Exclusion Criteria:

* Diabetes
* Overt cardiovascular disease
* Raynauds disease
* Current treatment with any anti-hypertensive, oral hypoglycaemic or lipid lowering therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-05; Primary Completion 2014-08-01 (Actual); Study Completion 2014-08-01 (Actual)

PRIMARY OUTCOMES:
Capillary pressure | 3 months
  Capillary pressure will be reduced in those treated with DPP-4 inhibitor

SECONDARY OUTCOMES:
Macular thickness | 3 months
  Measured by optical coherence tomography

CONTACTS AND LOCATIONS:
Locations (1):
- Diabetes and Vascular Research Department, Exeter, Devon, United Kingdom